CLINICAL TRIAL: NCT05293535
Title: Expression of Klotho and LRP-6 Proteins in Gastric Adenocarcinoma, is it an Important Issue??
Brief Title: Klotho _ LRP-6 _ Gastric Adenocarcinoma
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Collaborators: South Egypt Cancer Institute (Other)
Responsible Party: Principal Investigator, Marina Bassem Youssef Kostandy, Demonstator at Oncologic Pathology Department, South Egypt Cancer Institute, Assiut University, Assiut University
Other Study IDs: Klotho _ LRP-6 _ GC
Record Dates: First submitted 2022-03-11; First posted 2022-03-24 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Gastric Adenocarcinoma; Klotho; LRP-6

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Klotho: Evaluate the expression of Klotho in gastric adenocarcinoma via immunohistochemistry, find the association between the expression of Klotho in gastric adenocarcinoma and demographic patient data, and clinicopathologic parameters of the patients and investigate the effect of Klotho expression on the prognosis of gastric adenocarcinoma.
  Correlate between the Klotho and LRP-6 protein expression.
  Interventions: Other: Prognostic study
- LRP-6: Evaluate the expression of LRP-6 protein in gastric adenocarcinoma via immunohistochemistry, find the association between the expression of LRP-6 protein in gastric adenocarcinoma and demographic patient data, and clinicopathologic parameters of the patients and investigate the effect of LRP-6 protein expression on the prognosis of gastric adenocarcinoma.
  Correlate between the Klotho and LRP-6 protein expression.
  Interventions: Other: Prognostic study

INTERVENTIONS:
Other: Prognostic study — No intervention... as it is a prognostic study and no intervention done on patients.

SUMMARY:
Gastric cancer is the fifth most common malignancy in the world after cancers of the lung, breast, colorectum, and prostate. Gastric cancer is the third leading cause of cancer death and is responsible for 723,000 deaths yearly. Gastric carcinoma (GC) is a multifactorial disease which is difficult to diagnose in early-stage because of a time lag between the onset of growth and the appearance of clinical presentation. So, its prognosis is poor as evidenced by the 5-year survival rate.

Klotho is anti-aging gene encoding a protein with multiple pleiotropic effect. Cancer and ageing share comparable principles.

Klotho gene has been described as a tumor suppressor gene in numerous solid tumors and hematological malignancies. Klotho expression has been shown to be significantly down-regulated in malignant tissue compared to adjacent non-malignant tissue with good prognosis in cancers with high Klotho expression, including colorectal, pancreatic, gastric, esophageal, breast, hepatocellular, ovarian, and renal carcinomas. In contrast, a recent study documented that Klotho negative invasive duct carcinoma group exhibited good prognosis than the Klotho positive group regarding the disease- free survival after the surgical resection in breast cancer patient.

Lipoprotein receptor- related protein 6 (LRP6) is a type I single transmembrane protein which is a member of the low-density lipoprotein receptor (LDLR) gene family of receptors that is highly conserved among species. In 2000, LRP6 was identified as a co-receptor for Wnt and Frizzled (FZD) to transduce Wnt/β-catenin signaling. Dysregulation of LRP6 is involved in cancer. LRP6 is highly expressed in several cancer cell lines and overexpression of LRP6 promotes cancer cell proliferation. LRP6 expression is frequently upregulated in breast cancer tissue, and respective overexpression or knockdown of LRP6 induces or inhibits breast tumorigenesis. LRP6 is highly expressed in tumors of liver cancer patients, and overexpression of LRP6 promotes liver cancer cell proliferation and tumor growth. In prostate cancer, high expression levels of LRP6 are detected which activate Wnt/β-catenin signaling and glycolysis through Akt signaling. The end result is increased prostate cancer cell proliferation.

The mechanism of Klotho-mediated Wnt inhibition was as a result of Klotho binding to Wnt ligands, namely Wnt3A and Wnt5A; thereby impeding binding of these ligands to their cell surface receptor.

DETAILED DESCRIPTION:
Gastric cancer is the fifth most common malignancy in the world after cancers of the lung, breast, colorectum, and prostate. Gastric cancer is the third leading cause of cancer death and is responsible for 723,000 deaths yearly [1]. Gastric carcinoma (GC) is a multifactorial disease, where many factors can influence its development, both genetic and environmental such as infection with Helicobacter pylori (which is the main risk factor), gastric ulcer disease, gastroesophageal reflux disease and obesity [2]. Furthermore, genetic variations in proinflammatory and anti-inflammatory cytokine genes also influence the individual response to carcinogenic exposures. Host genetic factors are emerging as key determinants of disease risk for many cancers [1].

Gastric carcinoma is difficult to diagnose in early-stage because of a time lag between the onset of growth and the appearance of clinical presentation. Early symptoms of gastric cancer are not specific; as a result, most patients with early gastric cancer present with symptoms indistinguishable from benign peptic ulcer disease and, subsequently, these patients have been diagnosed at an advanced stage GC [1]. So, its prognosis is poor as evidenced by the 5-year survival rate and because most cases are already metastatic when diagnosed [2]. GC mostly affects older people. The average age of people when they are diagnosed with gastric cancer is 68 years [1].

Klotho is anti-aging gene encoding a protein with multiple pleiotropic effects, discovered in 1997 by Kuro-o and colleagues. The Klotho family of proteins consists of three members: α-Klotho, β-Klotho and γ-Klotho. All three are single-pass transmembrane proteins. The α-Klotho gene is composed of five exons, in humans, mice and rats expressed predominantly in the distal convoluted tubule (DCT) cells of the kidney in addition to a lesser expression in the proximal convoluted tubule (PCT) cells [3].

Cancer and ageing share comparable principles; the time-dependent accumulation of DNA damage is a contributing factor in ageing and also drives cancer progression. DNA damage, alongside genomic instability, is an established hallmark of most cancers. These pathways influence a number of capabilities acquired by cancer cells including the ability to evade apoptosis, cause tumor invasion and metastasis, sustain angiogenesis, and facilitate unlimited cellular replicative potential. Alpha-Klotho potentially influences these phenotypes through the inhibition of a number of signaling pathways such as insulin-like growth factor 1 receptor (IGF-1R), fibroblast growth factor (FGF), transforming growth factor β (TGFβ) and wingless-related integration site (Wnt) [4].

Klotho gene has been described as a tumor suppressor gene in numerous solid tumors and hematological malignancies, Klotho represents a possible therapeutic target for patients with these diseases, the majority of whom have limited treatment options [5].

Klotho expression has been shown to be significantly down-regulated in malignant tissue compared to adjacent non-malignant tissue with good prognosis in cancers with high Klotho expression, including colorectal [6], pancreatic [7], gastric [8], esophageal [9], breast [10], hepatocellular [11], ovarian [12], and renal carcinomas [13]. In contrast, a recent study done by Suzuki et al, 2021 documented that Klotho negative invasive duct carcinoma group exhibited good prognosis than the Klotho positive group regarding the disease- free survival after the surgical resection in breast cancer patient [14].

Lipoprotein receptor- related protein 6 (LRP6) is a type I single transmembrane protein which is a member of the low-density lipoprotein receptor (LDLR) gene family of receptors that is highly conserved among species. In 2000, LRP6 was identified as a co-receptor for Wnt and Frizzled (FZD) to transduce Wnt/β-catenin signaling. The extracellular domain of LRP6 interacts with Wnt and activates Wnt/β-catenin signaling at the plasma membrane. LRP6 with a truncated extracellular domain is constitutively active and can potentiate Wnt/β-catenin signaling independently of Wnt. Dysregulation of LRP6 is involved in cancer. LRP6 is highly expressed in several cancer cell lines and overexpression of LRP6 promotes cancer cell proliferation [15].

LRP6 expression is frequently upregulated in breast cancer tissue, and respective overexpression or knockdown of LRP6 induces or inhibits breast tumorigenesis [16]. LRP6 is highly expressed in tumors of liver cancer patients, and overexpression of LRP6 promotes liver cancer cell proliferation and tumor growth [17]. In prostate cancer, high expression levels of LRP6 are detected which activate Wnt/β-catenin signaling and glycolysis through Akt signaling. The end result is increased prostate cancer cell proliferation [19].

The mechanism of Klotho-mediated Wnt inhibition was as a result of Klotho binding to Wnt ligands, namely Wnt3A and Wnt5A; thereby impeding binding of these ligands to their cell surface receptor [4].

Klotho has also been shown to increase the efficacy of chemotherapy, including cisplatin in human lung cancer by modulating the phosphatidylinositol 3-kinase/protein kinase B PI3K/Akt pathway, indicating that Klotho therapy may be effective in combination with existing cancer therapies [4].

To our knowledge, it is the first research to study the expression of Klotho and LRP-6 protein in gastric adenocarcinoma by immunohistochemistry.

ELIGIBILITY:
Inclusion Criteria:

* Patients had a pathological diagnosis of gastric adenocarcinoma.
* Staging, lymph node (LN) metastasis and overall survival (OS) were analyzed according to Klotho and LRP-6 expression status.

Exclusion Criteria:

* Gastric Tumors other than adenocarcinoma.
* Cases with loss records files.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study is retrospective cohort study of 40-50 cases of gastric adenocarcinoma in our South Egypt Cancer Institute in the period from 2016 to 2020.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Expression of Klotho and LRP-6 proteins in gastric adenocarcinoma | 1-2 years
  Expression of Klotho and LRP-6 proteins in gastric adenocarcinoma via immunohistochemistry.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wong MCS, Huang J, Chan PSF, Choi P, Lao XQ, Chan SM, Teoh A, Liang P. Global Incidence and Mortality of Gastric Cancer, 1980-2018. JAMA Netw Open. 2021 Jul 1;4(7):e2118457. doi: 10.1001/jamanetworkopen.2021.18457. PMID 34309666
- [Background] Dermaku-Sopjani M, Kolgeci S, Abazi S, Sopjani M. Significance of the anti-aging protein Klotho. Mol Membr Biol. 2013 Dec;30(8):369-85. doi: 10.3109/09687688.2013.837518. Epub 2013 Oct 14. PMID 24124751
- [Background] Zhou X, Fang X, Jiang Y, Geng L, Li X, Li Y, Lu K, Li P, Lv X, Wang X. Klotho, an anti-aging gene, acts as a tumor suppressor and inhibitor of IGF-1R signaling in diffuse large B cell lymphoma. J Hematol Oncol. 2017 Feb 2;10(1):37. doi: 10.1186/s13045-017-0391-5. PMID 28153033
- [Background] Li XX, Huang LY, Peng JJ, Liang L, Shi DB, Zheng HT, Cai SJ. Klotho suppresses growth and invasion of colon cancer cells through inhibition of IGF1R-mediated PI3K/AKT pathway. Int J Oncol. 2014 Aug;45(2):611-8. doi: 10.3892/ijo.2014.2430. Epub 2014 May 9. PMID 24818842
- [Background] Jiang B, Gu Y, Chen Y. Identification of novel predictive markers for the prognosis of pancreatic ductal adenocarcinoma. Cancer Invest. 2014 Jul;32(6):218-25. doi: 10.3109/07357907.2014.905586. Epub 2014 Apr 18. PMID 24745611
- [Background] Wang L, Wang X, Wang X, Jie P, Lu H, Zhang S, Lin X, Lam EK, Cui Y, Yu J, Jin H. Klotho is silenced through promoter hypermethylation in gastric cancer. Am J Cancer Res. 2011;1(1):111-119. Epub 2010 Nov 10. PMID 21969138
- [Background] Tang X, Fan Z, Wang Y, Ji G, Wang M, Lin J, Huang S. Expression of klotho and beta-catenin in esophageal squamous cell carcinoma, and their clinicopathological and prognostic significance. Dis Esophagus. 2016 Apr;29(3):207-14. doi: 10.1111/dote.12289. Epub 2014 Oct 6. PMID 25287007
- [Background] Wolf I, Levanon-Cohen S, Bose S, Ligumsky H, Sredni B, Kanety H, Kuro-o M, Karlan B, Kaufman B, Koeffler HP, Rubinek T. Klotho: a tumor suppressor and a modulator of the IGF-1 and FGF pathways in human breast cancer. Oncogene. 2008 Nov 27;27(56):7094-105. doi: 10.1038/onc.2008.292. Epub 2008 Sep 1. PMID 18762812
- [Background] Tang X, Wang Y, Fan Z, Ji G, Wang M, Lin J, Huang S, Meltzer SJ. Klotho: a tumor suppressor and modulator of the Wnt/beta-catenin pathway in human hepatocellular carcinoma. Lab Invest. 2016 Feb;96(2):197-205. doi: 10.1038/labinvest.2015.86. Epub 2015 Aug 3. PMID 26237271
- [Background] Yan Y, Wang Y, Xiong Y, Lin X, Zhou P, Chen Z. Reduced Klotho expression contributes to poor survival rates in human patients with ovarian cancer, and overexpression of Klotho inhibits the progression of ovarian cancer partly via the inhibition of systemic inflammation in nude mice. Mol Med Rep. 2017 Apr;15(4):1777-1785. doi: 10.3892/mmr.2017.6172. Epub 2017 Feb 7. PMID 28259911
- [Background] Gigante M, Lucarelli G, Divella C, Netti GS, Pontrelli P, Cafiero C, Grandaliano G, Castellano G, Rutigliano M, Stallone G, Bettocchi C, Ditonno P, Gesualdo L, Battaglia M, Ranieri E. Soluble Serum alphaKlotho Is a Potential Predictive Marker of Disease Progression in Clear Cell Renal Cell Carcinoma. Medicine (Baltimore). 2015 Nov;94(45):e1917. doi: 10.1097/MD.0000000000001917. PMID 26559258
- [Background] Suzuki S, Sakurai K, Hirano T, Adachi K, Koshinaga T, Makishima M. [Prediction of Prognosis in Breast Carcinoma Using Klotho Immunohistochemistry]. Gan To Kagaku Ryoho. 2021 Aug;48(8):1043-1047. Japanese. PMID 34404073
- [Background] Jeong W, Jho EH. Regulation of the Low-Density Lipoprotein Receptor-Related Protein LRP6 and Its Association With Disease: Wnt/beta-Catenin Signaling and Beyond. Front Cell Dev Biol. 2021 Sep 13;9:714330. doi: 10.3389/fcell.2021.714330. eCollection 2021. PMID 34589484
- [Background] Zhang J, Li Y, Liu Q, Lu W, Bu G. Wnt signaling activation and mammary gland hyperplasia in MMTV-LRP6 transgenic mice: implication for breast cancer tumorigenesis. Oncogene. 2010 Jan 28;29(4):539-49. doi: 10.1038/onc.2009.339. Epub 2009 Nov 2. PMID 19881541
- [Background] Tung EK, Wong BY, Yau TO, Ng IO. Upregulation of the Wnt co-receptor LRP6 promotes hepatocarcinogenesis and enhances cell invasion. PLoS One. 2012;7(5):e36565. doi: 10.1371/journal.pone.0036565. Epub 2012 May 3. PMID 22570728
- [Background] Lemieux E, Cagnol S, Beaudry K, Carrier J, Rivard N. Oncogenic KRAS signalling promotes the Wnt/beta-catenin pathway through LRP6 in colorectal cancer. Oncogene. 2015 Sep 17;34(38):4914-27. doi: 10.1038/onc.2014.416. Epub 2014 Dec 15. PMID 25500543
- [Background] Tahir SA, Yang G, Goltsov A, Song KD, Ren C, Wang J, Chang W, Thompson TC. Caveolin-1-LRP6 signaling module stimulates aerobic glycolysis in prostate cancer. Cancer Res. 2013 Mar 15;73(6):1900-11. doi: 10.1158/0008-5472.CAN-12-3040. Epub 2013 Jan 9. PMID 23302227
- [Background] Liu H, Fergusson MM, Castilho RM, Liu J, Cao L, Chen J, Malide D, Rovira II, Schimel D, Kuo CJ, Gutkind JS, Hwang PM, Finkel T. Augmented Wnt signaling in a mammalian model of accelerated aging. Science. 2007 Aug 10;317(5839):803-6. doi: 10.1126/science.1143578. PMID 17690294